CLINICAL TRIAL: NCT04087837
Title: Using Bougie or Cooled Nasogastric Tube to Facilitate Nasotracheal Tube Advancement Into Trachea Under Video-laryngoscope
Brief Title: The Effectiveness of Using Bougie or Cooled Nasogastric Tube to Facilitate Nasotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pin-Yang Hu, MD, physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20190075
Record Dates: First submitted 2019-09-01; First posted 2019-09-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Intubation Complication
Keywords: bougie, nasotracheal tube; Endotracheal Tube intubation General Anesthesia (ETGA)

STUDY DESIGN:
Intervention Model Description: bougie or nasogastric tube
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bougie group (Experimental): The bougie group: The end of the endotracheal tube was guided to the glottis using the endotracheal tube in the bougie mode under the direct view of the electronic imaging laryngoscope. The Magill Forceps is used to assist the tip of the endotracheal tube in guiding the glottis.
  Interventions: Device: bougie
- Nasogastric(NG) tube group (Experimental): NG tube group: The end of the endotracheal tube is guided to the glottis by using the endotracheal tube in the nasogastric tube under the direct view of the electronic imaging laryngoscope. The Magill Forceps is used to assist the tip of the endotracheal tube in guiding the glottis.
  Interventions: Device: Nasogastric(NG) tube
- control group (No Intervention): Control group: The general anesthesia method of placing the endotracheal tube through the nasal cavity is used to guide the tip of the endotracheal tube to the glottis under the direct view of the electronic imaging laryngoscope.

INTERVENTIONS:
Device: bougie — The endotracheal tube is used in the bougie mode under the direct view of the electronic imaging laryngoscope.
  Arms: bougie group
Device: Nasogastric(NG) tube — The endotracheal tube is used in the NG tube mode under the direct view of the electronic imaging laryngoscope.
  Arms: Nasogastric(NG) tube group

SUMMARY:
either uses a bougie or nasogastric tube to assist the nasotracheal tube passing the nasal cavity, nasopharynx, oropharynx and advanced into the trachea

DETAILED DESCRIPTION:
In oro-maxillo-facial surgery, it is a common practice for patients receiving general anesthesia with nasotracheal intubation to widen the surgical field and to ease undergoing surgery. However, a nasotracheal tube blindly passing through the nasal cavity may easily result in nasal cavity and oropharynx damages. In addition, the advancement of the tube from oropharynx into trachea may assist by either using magic forceps or cuff inflation technique.

The aim of the study is to investigate either use a bougie or nasogastric tube to assist the nasotracheal tube passing the nasal cavity, nasopharynx, oropharynx, and advanced into the trachea.

Patients were randomized into three groups by using either bougie or nasogastric tube to facilitate nasotracheal tube sliding through into trachea from assigned nostril and compared with the control group with a conventional technique.

Hemodynamic changes in each time interval, each time taken of tube going through the nasal cavity, tube advanced from oropharynx into trachea were recorded. The incidence of using Magill Forceps to accurately place tube tip into trachea, intubation related side effects and complications were recorded at postoperative time stages.

ELIGIBILITY:
Inclusion Criteria:

* Age:20-65 years
* Undergoing oro-maxillofacial surgery
* Opening mouth > 3 cm
* Denied any systemic disease.
* American Society of Anesthesiologists (ASA) class:I-III

Exclusion Criteria:

* Difficult airway assessed (limited mouth opening, limited neck motion, and thyromental distance < 6cm)
* Previous head and neck surgery history
* Upper abnormal airway diagnosed
* Easily epistaxis
* Both sides nasal cavities obstruction

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
success rate of tube advancement and successful first tube attempt | 10 minutes
  success rate of tube passing through nasal cavity into trachea
time taken in tube advancement | 10 minutes
  time taken in tube advancement from nostril into trachea in each time interval

SECONDARY OUTCOMES:
post-intubation induced hoarseness and sore throat | 2 days
  A visiting questionnaire is used to measure the condition of post-intubation, including sore throat, hoarseness, dysphagia, nasal occlusion, nosebleed and nasal pain. The score for the measurement of sore throat, hoarseness, dysphagia is divided into four degrees: none, mild, moderate and severe; on the other hand, The score for the measurement of nasal occlusion, nosebleed and nasal pain is divided into yes or no. All the evaluation will be assessed in the next coming morning after the postoperation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesiology, Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan